CLINICAL TRIAL: NCT03412227
Title: Randomized Clinical Trial of Transdiagnostic Behavioral Activation and Exposure Therapy for Youth: A Comparison of Effects and Mediators
Brief Title: Transdiagnostic Individual Behavioral Activation and Exposure Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Brian C. Chu, Associate Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro20170001171
Record Dates: First submitted 2017-10-15; First posted 2018-01-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Disorders; Depression
Keywords: Anxiety; Depression; Children; Adolescents; CBT
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial, stratified by principal youth diagnosis (anxiety or depression).
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be masked to the treatment conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Principal Anxiety Disorder (Other): Youth with a principal anxiety disorder
  Interventions: Behavioral: Individual Behavioral Activation Therapy (IBAT); Behavioral: The Coping Cat Program for Youth Anxiety Disorders; Other: 14-week waitlist (WL) condition
- Principal Depressive Disorder (Other): Youth with a principal unipolar depressive disorder
  Interventions: Behavioral: Individual Behavioral Activation Therapy (IBAT); Behavioral: The PASCET Program for Youth Depressive Disorders; Other: 14-week waitlist (WL) condition

INTERVENTIONS:
Behavioral: Individual Behavioral Activation Therapy (IBAT) — IBAT is a manual-based, individual behavioral activation plus exposure therapy aimed at treating youth with anxiety, depression, and anger. The program consists of 10-14 weekly 60 minute sessions. It uses behavioral activation (BA) strategies to target avoidance by helping youth identify stuck points in their lives through functional assessment of numerous life domains, including family and peer interactions, school, extracurricular activities, and health and self-care.
Behavioral: The PASCET Program for Youth Depressive Disorders — The Primary and Secondary Control Enhancement Therapy (PASCET; Weisz, Southam-Gerow, Gordis, & Connor-Smith, 2003; Weisz, Southam-Gerow et al., 2009; Weisz, Thurber, Sweeney, Proffitt, & LeGagnoux, 1997) is a brief (usually 11-15 sessions) CBT program for depressed youths typically aged 8-15. Sessions and practice assignments are built on findings concerning cognitive and behavioral features of, and beneficial treatments for, youth depression (e.g., Lewinsohn et al., 1990; Stark et al., 1987), and on the two-process model of perceived control and coping (Rothbaum, Weisz, & Snyder, 1982; Weisz et al., 1984a,b).
  Arms: Principal Depressive Disorder
Behavioral: The Coping Cat Program for Youth Anxiety Disorders — The "Coping Cat" program (Kendall & Hedtke, 2006; Kendall, Choudhury, Hudson, & Webb, 2002) has received substantial empirical support for its efficacy in both children (9-13 years old) and teens (12 - 17 years old) (Kendall, 1994; Kendall et al., 1997; Kendall et al., 2008) and involves (1) teaching children to identify their own anxious feelings and physiological signs of anxiety, (2) teaching children to identify their own anxiety-provoking cognitions, (3) developing a plan to guide coping - a plan that involves changing the child's thoughts (into positive self-talk) and actions (into self-initiated exposures), and (4) self-evaluation and self-reward.
  Arms: Principal Anxiety Disorder
Other: 14-week waitlist (WL) condition — Youth assigned to the 14-week WL will receive no specific therapeutic services from study therapists during the 14-week WL period. However, participants will be assigned a WL Liaison whom families can contact in the event of clinical deterioration. The Liaison will also be responsible for sending links to, and monitor completion of, weekly and mid-WL online surveys (Qualtrics). Independent Evaluators will conduct post-WL diagnostic interviews at the completion of the 14-week WL. WL participants will receive compensation for completion of assessments. After completion of the WL, participants will be invited to continue in the study and be randomly assigned to one of the three behavioral treatments (IBAT, PASCET, or Coping Cat).

SUMMARY:
The Overall Aim of the this project is to compare treatment outcomes and change in putative treatment mediators in Individual Behavioral Activation Therapy (IBAT) against two active psychological interventions (Coping Cat, PASCET) and a wait-list control. Participants will be 200 youth (ages 9-17) diagnosed with a principal anxiety or depression disorder and their caregivers.

DETAILED DESCRIPTION:
Anxiety and unipolar depression are highly debilitating and commonly co-occurring in young adolescents with lifetime prevalence rates estimated at 8.4% for major depression or dysthymia and at 31.4% for any anxiety disorder in youth ages 13-14 (Merikangas et al., 2010). Cognitive and behavioral therapies (CBT) have received strong support for reducing distress in youth (Silverman, Pina, & Viswesvaran, 2008; David-Ferdon & Kaslow, 2008), but efficacy rates peak around 50-70% for anxiety and less for depression. Evidence is accumulating that "transdiagnostic" behavioral therapies that address multiple problems at the same time can enhance treatment outcomes by targeting the mechanisms that underlie commonly co-occurring problems, like anxiety and depression (Chu, Temkin, & Toffey, 2016; Temkin, Yadegar, Laurine, & Chu, in press). Furthermore, consolidated transdiagnostic treatment protocols can provide the same level of clinical benefit while delivering active components in a more efficient package, which can increase treatment efficiency and potentially make it easier to train novice clinicians in the future (Chu, 2012; Ehrenreich & Chu, 2013). While the evidence-base is growing for adult conditions, transdiagnostic interventions have been examined less in child and adolescent populations. Our team has demonstrated the efficacy of a school-based group transdiagnostic intervention that made use of behavioral activation (BA) and exposure therapy to address anxiety and depression for middle-school youth (Chu, Crocco, Esseling, Areizaga, Lindner, & Skriner, 2016). BA refers to a set of interventions that teach youth how to assess which stressors trigger avoidant coping responses in their lives (i.e., functional assessment) and learn how to address problems with pro-active problem solving strategies. Exposure therapy refers to a set of behavioral interventions that foster new learning tendencies by encouraging and reinforcing contact with the situations that scare individuals. Both sets of strategies have received substantial support in treating youth anxiety and depression. The Chu et al., (2016) trial demonstrated that these two treatment components could be combined and effectively treat a sample of youth reporting either anxiety or depression.

The Chu et al. (2016) study was novel because most forms of evidence-based treatment have been designed as "single disorder" protocols, such that the interventions were designed to target one clinical problem at a time. The current trial takes the following innovative steps. The study will: (a) adapt the Chu et al. group-based protocol to an individual format, (b) deliver the program in a clinical outpatient setting, and (c) utilize three comparison conditions, including a wait-list control and two active psychological interventions. The two active interventions will be single disorder cognitive behavioral therapies (CBT) that were designed to specifically address either youth depression (Primary and Secondary Control Enhancement Therapy; PASCET; Weisz, Thurber, Sweeney, Proffitt, & LeGagnoux, 1997) or youth anxiety (Coping Cat; Kendall, 1994; Kendall et al., 1997). Both have received substantial support in the literature for supporting clinical improvements in brief individual formats (12 - 16 weeks). By comparing Individual Behavioral Activation Therapy (IBAT) to each of these active interventions, the study aims to demonstrate (a) superior treatment outcomes to wait-list control, (b) comparable treatment outcomes to PASCET and Coping Cat, and (c) differential mediator effects across the four conditions. Findings will provide support for the feasibility, acceptability, and efficacy of IBAT and provide conceptual support for its purported mediators of change.

The current study is a Randomized Controlled Trial (RCT), comparing a novel behavioral intervention (Individual Behavioral Activation Therapy, IBAT) against two established cognitive-behavioral interventions (Coping Cat, PASCET) and a 14-week waitlist (WL) control. Participants will be 160 youth (ages 9-16 years old) who receive a diagnosis of a Diagnostic and Statistical Manual - 5th edition (DSM-5; APA, 2013) anxiety or depression disorder and their caregivers. Participants will be randomly assigned evenly to each of four conditions. The study intends to recruit participants within a 2.5-year period and complete all active participant participation within 3 years.

Specific aims include the following:

Aim 1 - Treatment Efficacy: To evaluate differences in treatment outcomes across IBAT, PASCET, CC, and WL conditions across pre-, mid-, and post-treatment in treatment efficacy, focusing on key diagnostic and symptom outcomes (i.e., CGI, principal diagnosis presence to absence and clinical severity, RCADS anxiety and depression scores, MASC, CESD).

Hypothesis 1: IBAT will produce superior outcomes to 14-week WL control

Hypothesis 2: The three active treatment conditions (IBAT, PASCET, CC) will demonstrate superior treatment outcomes to 14-week WL control, but will not be different from each other.

Aim 2 - Mediator Analysis: To examine the strength of putative mediators in explaining the effects of active treatments (IBAT, CC, PASCET) in comparison to the 14-week WL and in comparison to each other. Putative mediators will include multiple domains: (a) youth socio-emotional functioning (cognitive, behavioral, and affective responses), (b) distress tolerance as assessed by computer tasks, (c) family environment and interactions, (d) caregiver distress and functioning, (e) client and therapist perception of psychotherapy process, (f) ecological momentary assessment and passive sensor data.

Hypothesis 3: Each domain will prove to provide significant mediators for each treatment in comparison to the WL control.

Hypothesis 4: Cognitive mediators will prove to provide significant mediation of CC and PASCET treatment effects, but not necessarily for IBAT.

Hypothesis 5: Distress tolerance will prove to provide significant mediator for IBAT treatment effects, but not necessarily for CC or PASCET.

Aim 3. Note patterns of additional youth mental health services and auxiliary services that families seek beyond treatment received at the Youth Anxiety and Depression Clinic.

ELIGIBILITY:
We expect 200 youth (ages 9-17 years) with either a principle anxiety (n=100) or a unipolar depression disorder (n=100) and their parents/caregivers to serve as participants.

Inclusion Criteria:

To participate, a youth must meet criteria for a primary DSM-5 (American Psychiatric Association, 2003) diagnosis of any of the following:

* Generalized Anxiety Disorder (GAD)
* Separation Anxiety Disorder (SEP)
* Social Anxiety Disorder (SAD)
* Specific Phobia (SP)
* Panic Disorder (PD)
* Agoraphobia
* Major Depression Disorder (MDD)
* Depression Disorder - Insufficient Symptoms (DD-Insufficient)
* Persistent Depressive Disorder (PDD)

Comorbid (non-principal) disorders are acceptable, including the presence of disorders not listed above. Diagnosis will be based on both youth and parent report during an Independent Evaluator (IE) semi-structured interview. Youth may also participate with a subclinical diagnosis for any of these disorders if: (a) the youth demonstrates sufficient symptoms but does not yet reach clinical levels of impairment OR (b) the youth demonstrates only several symptoms related to the above disorders but demonstrates clinical impairment, AND (c) the consenting parent agrees that anxiety or mood problems would be appropriate as a clinical focus for treatment. Allowing youth with subclinical diagnoses will allow the study to investigate the effectiveness of the therapies across a range of clinical severity. This design models usual community care where a larger range of severity is witnessed and many youth may not meet all criteria for formal diagnosis. After receiving an initial diagnostic assessment at T1, the parent must consent and the youth must assent to continued participation in the study, including randomization to treatment condition, and must be willing to receive psychological therapy at the Youth Anxiety and Depression Clinic (YAD-C), a specialty program within the outpatient clinic of the Rutgers University Graduate School of Applied and Professional Psychology (GSAPP).

Exclusion Criteria:

Youth who have a principal DSM-5 disorder other than one of the above listed anxiety or depression disorders (e.g., anorexia nervosa, Post-traumatic Stress Disorder, Attention Deficit-Hyperactivity Disorder), or who have received any diagnosis of:

* Intellectual Disability
* Autism Spectrum Disorder
* schizophrenia
* bipolar disorder.

Youth who demonstrate suicidal ideation or intent (by child or parent report) severe enough to require current hospitalization, or youth who have attempted suicide in the past 3 months, will also be excluded. These clinical problems require specialized treatment that YAD-C is not prepared to offer. Youth will not be excluded on the basis of gender or racial/ethnic origin. However, youth and at least one parent will be required to speak English sufficiently enough to complete study procedures and surveys in English. Participants will be asked not to engage in any other outpatient psychological treatment during their time in the study; this is important to enhance internal validity of the study and conforms with best clinical practices to avoid conflicting treatment recommendations. However, current use of antidepressant or anxiolytic medications will NOT be an exclusion. Participants will be asked to arrive at a stable dosage and schedule for their medication, in consultation with their presiding physician or psychiatrist, prior to study initiation. Use of medications and any other treatment modalities will be assessed during study participation and compared across treatment and WL conditions.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression Severity (CGIS) Scale: Independent Evaluator | Change from pre-treatment to post-treatment (baseline to 14-weeks)
  The CGI-S score provides a global rating of baseline severity ranging from 1 (not at all ill) to 7 (extremely ill), while the CGI-I provides a global rating of clinical improvement ranging from 1 (Very Much Improved) to 7 (Very Much Worse). The IE will provide a baseline CGI ratings for each patient at pretreatment and posttreatment. Subjects receiving a CGI-I rating of 1 (Very Much Improved) or 2 (Much Improved) by the IE at the end of posttreatment will be considered responders of treatment.

SECONDARY OUTCOMES:
Change in Behavioral Activation | Change from pre-treatment to post-treatment (baseline to 14-weeks)
  The BADS-Y is a 26-item adaptation of the adult BADS (Kanter et al., 1997; Kanter et al., 1999), rated on a "0" (Not at All) to "6" (Completely) scale, designed to assess level of behavioral activation and avoidance. Factor analysis in the adult version detected four factors: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment) with good factor structure, internal consistency and test-retest reliability. Normative data was also collected in an adult community sample. BADS-A was adapted for the current study to reflect developmentally appropriate reading level and concepts.
Child Automatic Thoughts Scale-Negative/Positive | Change from pre-treatment to post-treatment (baseline to 14-weeks)
  The CATS is a 50-item child-report measure designed to assess negative and positive self-statements in children and adolescents. The CATS was developed and validated on a wide age range of youth (7 - 16 years old) and found to effectively discriminate between non-clinical youth and those with clinical anxiety, depression, and behavior disorders. Confirmatory factor analyses supported four distinct but strongly correlated factors relating to automatic thoughts on physical threat, social threat, personal failure and hostility. The internal consistency of the total score and subscales was high (α > .85) and test-retest reliability at 1 and 3 months was acceptable (r = .91).

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Chu, Ph.D., Principal Investigator — Rutgers University (Youth Anxiety and Depression Clinic)
Locations (1):
- Youth Anxiety and Depression Clinic, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GenIUSS (2014). Best practices for asking questions to identify transgender and other gender minority respondents on population-based surveys. Retrieved from https://williamsinstitute.law.ucla.edu/wp-content/uploads/geniuss-report-sep-2014.pdf
- [Background] Fenway Institute (n.d.). Asking patients questions about sexual orientation and gender identity in clinical settings: A study in four health centers. Retrieved from http://thefenwayinstitute.org/wp-content/uploads/COM228_SOGI_CHARN_WhitePaper.pdf
- [Background] Official New York City Website (n.d.). Respectfully asking sexual orientation and gender identity (SOGI) questions. Retrieved from https://www1.nyc.gov/assets/acs/pdf/lgbtq/Respectfully_Asking_SOGI_Questions.pdf
- [Background] Achenbach, T. M. (2001). Manual for the ASEBA Child Behavior Checklist for Ages 6-18. Burlington, VT: Achenbach System of Empirically Based Assessment.
- [Background] American Psychiatric Association (2000). Diagnostic and Statistical Manual of Mental Disorders-IV-TR (4th Ed., Text Revision). Arlington, VA: American Psychiatric Association.
- [Background] American Psychiatric Association (2013). Diagnostic and Statistical Manual of Mental Disorders-IV-TR (5th Ed.). Arlington, VA: American Psychiatric Association.
- [Background] Ashrafioun L, Dambra CM, Blondell RD. Parental prescription opioid abuse and the impact on children. Am J Drug Alcohol Abuse. 2011 Nov;37(6):532-6. doi: 10.3109/00952990.2011.600387. Epub 2011 Aug 18. PMID 21851201
- [Background] Barlow, D. H. & Hersen, M. (1984). Single-case experimental designs: Strategies for studying behavior change (2nd Ed.). New York: Pergamon Press.
- [Background] Barrett PM, Rapee RM, Dadds MM, Ryan SM. Family enhancement of cognitive style in anxious and aggressive children. J Abnorm Child Psychol. 1996 Apr;24(2):187-203. doi: 10.1007/BF01441484. PMID 8743244
- [Background] Bornovalova MA, Gratz KL, Daughters SB, Nick B, Delany-Brumsey A, Lynch TR, Kosson D, Lejuez CW. A multimodal assessment of the relationship between emotion dysregulation and borderline personality disorder among inner-city substance users in residential treatment. J Psychiatr Res. 2008 Jul;42(9):717-26. doi: 10.1016/j.jpsychires.2007.07.014. Epub 2007 Sep 14. PMID 17868698
- [Background] Brandon TH, Herzog TA, Juliano LM, Irvin JE, Lazev AB, Simmons VN. Pretreatment task persistence predicts smoking cessation outcome. J Abnorm Psychol. 2003 Aug;112(3):448-56. doi: 10.1037/0021-843x.112.3.448. PMID 12943023
- [Background] Carey MP, Faulstich ME, Carey TC. Assessment of anxiety in adolescents: concurrent and factorial validities of the Trait Anxiety scale of Spielberger's State-Trait Anxiety Inventory for Children. Psychol Rep. 1994 Aug;75(1 Pt 1):331-8. PMID 7984747
- [Background] Chorpita BF, Weisz JR, Daleiden EL, Schoenwald SK, Palinkas LA, Miranda J, Higa-McMillan CK, Nakamura BJ, Austin AA, Borntrager CF, Ward A, Wells KC, Gibbons RD; Research Network on Youth Mental Health. Long-term outcomes for the Child STEPs randomized effectiveness trial: a comparison of modular and standard treatment designs with usual care. J Consult Clin Psychol. 2013 Dec;81(6):999-1009. doi: 10.1037/a0034200. Epub 2013 Aug 26. PMID 23978169
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Chu BC, Kendall PC. Therapist responsiveness to child engagement: flexibility within manual-based CBT for anxious youth. J Clin Psychol. 2009 Jul;65(7):736-54. doi: 10.1002/jclp.20582. PMID 19391153
- [Background] Chu, B. C. (2012). Introduction to special series: Translating transdiagnostic approaches to children and adolescents. Cognitive and Behavioral Practice, 19, 1-4.
- [Background] Chu, B. C., Colognori, D., Weissman, A. S., & Bannon, K. (2009). An initial description and pilot of group behavioral activation therapy for anxious and depressed youth. Cognitive and Behavioral Practice, 16, 408-419.
- [Background] Chu BC, Crocco ST, Esseling P, Areizaga MJ, Lindner AM, Skriner LC. Transdiagnostic group behavioral activation and exposure therapy for youth anxiety and depression: Initial randomized controlled trial. Behav Res Ther. 2016 Jan;76:65-75. doi: 10.1016/j.brat.2015.11.005. Epub 2015 Nov 19. PMID 26655958
- [Background] Chu, B. C., Hoffman, L., Johns, A., Reyes-Portillo, J., & Hansford, A. (2015). Transdiagnostic behavior therapy for bullying-related anxiety and depression: Initial development and pilot study. Cognitive and Behavioral Practice, 22, 415-429. doi: 10.1016/j.cbpra.2014.06.007
- [Background] Chu, B. C., Merson, R. A., Zandberg, L. J., & Areizaga, M. (2012). Calibrating for comorbidity: Clinical decision-making in youth depression and anxiety. Cognitive and Behavioral Practice, 19, 5-16.
- [Background] Chu, B. C., Skriner, L. C., & Staples, A. M. (2013). Behavioral avoidance across anxiety, depression, impulse, and conduct problems. In J. Ehrenreich-May, & B. Chu, (Eds.), Transdiagnostic treatments for children and adolescents: Principles and practice (pp. 84 - 110). New York: Guilford Press.
- [Background] Chu, B. C., Temkin, A., & Toffey, K. (2016). Transdiagnostic mechanisms and treatment in child and adolescent research: An emerging field. In P. Nathan (Ed.), Oxford Handbooks Online. Downloaded Sept 7, 2016, from http://www.oxfordhandbooks.com/view/10.1093/oxfordhb/9780199935291.001.0001/oxfordhb-9780199935291-e-10. DOI: 10.1093/oxfordhb/9780199935291.013.10.
- [Background] Chorpita, B.F., Daleiden, E. L., Moffitt, C., Yim, L., & Umemoto, L. A. (2000). Assessment of tripartite factors of emotion in children and adolescent: I. Structural validity and normative data of an affect and arousal scale. Journal of Psychopathology and Behavioral Assessment, 22, 141-160.
- [Background] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Background] Connor, A., Franzen, M. D., & Sharp, B. (1988). Effects of practice and differential on Stroop performance. International Journal of Clinical Neuropsychology, 10, 1-4.
- [Background] Connor-Smith JK, Compas BE, Wadsworth ME, Thomsen AH, Saltzman H. Responses to stress in adolescence: measurement of coping and involuntary stress responses. J Consult Clin Psychol. 2000 Dec;68(6):976-92. PMID 11142550
- [Background] Costello, E. J. (1990). Child psychiatric epidemiology: Implications for clinical research and practice. In B. B. Lahey & A. E. Kazdin (Eds.), Advances in clinical child psychology (vol. 13, pp. 53-90). New York, NY: Plenum Press.
- [Background] Costello EJ. Developments in child psychiatric epidemiology. J Am Acad Child Adolesc Psychiatry. 1989 Nov;28(6):836-41. doi: 10.1097/00004583-198911000-00004. No abstract available. PMID 2681135
- [Background] Crosbie J. Interrupted time-series analysis with brief single-subject data. J Consult Clin Psychol. 1993 Dec;61(6):966-74. doi: 10.1037//0022-006x.61.6.966. PMID 8113497
- [Background] Dadds, M. R. & Barrett, P. M. (1996). Family processes in child and adolescent anxiety and depression. Behaviour Change, 13(4), 231-239.
- [Background] Dadds MR, Barrett PM, Rapee RM, Ryan S. Family process and child anxiety and aggression: an observational analysis. J Abnorm Child Psychol. 1996 Dec;24(6):715-34. doi: 10.1007/BF01664736. PMID 8970906
- [Background] Daleiden, E. L., Chorpita, B.F., & Lu, W. (2000). Assessment of tripartite factors of emotion in children and adolescent: II. Concurrent validity of the affect and arousal scales for children. Journal of Psychopathology and Behavioral Assessment, 22, 161-182.
- [Background] Daughters SB, Reynolds EK, MacPherson L, Kahler CW, Danielson CK, Zvolensky M, Lejuez CW. Distress tolerance and early adolescent externalizing and internalizing symptoms: the moderating role of gender and ethnicity. Behav Res Ther. 2009 Mar;47(3):198-205. doi: 10.1016/j.brat.2008.12.001. Epub 2008 Dec 13. PMID 19135649
- [Background] Digiuseppe, R., Linscott, J., & Jilton, R. (1996). Developing the therapeutic alliance in child-adolescent psychotherapy. Applied & Preventive Psychology, 5(2), 85-100.
- [Background] Ehrenreich-May, J. & Chu, B. C. (2013). Overview of transdiagnostic mechanisms and treatments for youth psychopathology. In J. Ehrenreich-May & B. C. Chu (Eds.), Transdiagnostic treatments for children and adolescents: Principles and practice (pp. 3-14). New York: Guilford Press.
- [Background] Finch AJ Jr, Kendall PC, Montgomery LE. Multidimensionality of anxiety in children. Factor structure of the Children's Manifest Anxiety Scale. J Abnorm Child Psychol. 1974 Dec;2(4):331-5. doi: 10.1007/BF00919262. No abstract available. PMID 4463193
- [Background] Gaynor, S. T., Baird, S. C., & Nelson-Gray, R. O. (1999). Application of time-series (single-subject) designs in clinical psychology. In P.C. Kendall, J.N. Butcher, & G.N. Holmbeck (Eds.), Handbook of research methods in clinical psychology, 2nd Ed. New York: John Wiley & Sons, Inc.
- [Background] Gioia G, Isquith P, Guy S, Kenworthy L (2000). BRIEF-Behavior Rating Inventory of Executive Function. Professional Manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Graf P, Uttl B, Tuokko H. Color- and picture-word Stroop tests: performance changes in old age. J Clin Exp Neuropsychol. 1995 May;17(3):390-415. doi: 10.1080/01688639508405132. PMID 7650102
- [Background] Guy, W. (1976). ECDEU Assessment Manual for Psychopharmacology (2nd ed.) (DHEW Publication ABM 76-388). Washington, DC: US Government Printing Office.
- [Background] Hankin BL, Gibb BE, Abela JR, Flory K. Selective attention to affective stimuli and clinical depression among youths: role of anxiety and specificity of emotion. J Abnorm Psychol. 2010 Aug;119(3):491-501. doi: 10.1037/a0019609. PMID 20677838
- [Background] Hawley, K., Weersing, V. R., & Weisz, J. R. (1998). Parent Child Satisfaction Scale. Unpublished Scale. Available from author.
- [Background] Hoagwood, K., Horwitz, S., Stiffman, A., Weisz, J., Bean, D., Rae, D., & ... Leaf, P. (2000). Concordance between parent reports of children's mental health services and service records: The Services Assessment for Children and Adolescents (SACA). Journal of Child and Family Studies, 9 (3), 315-331.
- [Background] Hodges, K. (1990). Depression and anxiety in children: A comparison of self-report questionnaires to clinical interview. Psychological Assessment, 2, 376-381.
- [Background] Horwitz SM, Hoagwood K, Stiffman AR, Summerfeld T, Weisz JR, Costello EJ, Rost K, Bean DL, Cottler L, Leaf PJ, Roper M, Norquist G. Reliability of the services assessment for children and adolescents. Psychiatr Serv. 2001 Aug;52(8):1088-94. doi: 10.1176/appi.ps.52.8.1088. PMID 11474056
- [Background] Holmbeck, G. N. Greenley, R. N., & Franks, E. A. (2003). Developmental issues and considerations in research and practice. In A. E. Kazdin & J. R. Weisz (Eds.), Evidence-based psychotherapies for children and adolescents (pp. 21-41). New York, NY: Guilford Press.
- [Background] Kanter, J. W., Mulick, P. S., Busch, A. M., Berlin, K. S., & Martell, C. R. (1997). The Behavioral Activation for Depression Scale (BADS): Psychometric properties and factor structure. Journal of Psychopathology Behavioral Assessment, 29, 191-202.
- [Background] Kanter, J. W., Rusch, L. C., Busch, A. M., & Sedivy, S. K. (1999). Validation of the Behavioral Activation for Depression Scale (BADS) in a community sample with elevated depressive symptoms. Journal of Psychopathology Behavioral Assessment, 31, 36-42.
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Kazdin AE, Weisz JR. Identifying and developing empirically supported child and adolescent treatments. J Consult Clin Psychol. 1998 Feb;66(1):19-36. doi: 10.1037//0022-006x.66.1.19. PMID 9489260
- [Background] Kazdin, A. E. (1992). Research Design in Clinical Psychology, 2nd Ed. Needham Heights, MA: Allyn & Bacon.
- [Background] Kendall PC. Treating anxiety disorders in children: results of a randomized clinical trial. J Consult Clin Psychol. 1994 Feb;62(1):100-10. doi: 10.1037//0022-006x.62.1.100. PMID 8034812
- [Background] Kendall, P. C., Aschenbrand, S. G., Hudson, J. L. (2003). Child-focused treatment of anxiety. In A. E. Kazdin & J. R. Weisz (Eds.), Evidence-based psychotherapies for children and adolescents (pp 81-100). New York, NY: Guilford Press.
- [Background] Kendall, P. C., Choudhury, M., Hudson, J., & Webb, A. (2002). The C.A.T. Project Manual for the Cognitive-behavioral treatment of anxious adolescents. Ardmore, PA: Workbook Publishing.
- [Background] Kendall PC, Flannery-Schroeder EC. Methodological issues in treatment research for anxiety disorders in youth. J Abnorm Child Psychol. 1998 Feb;26(1):27-38. doi: 10.1023/a:1022630706189. PMID 9566544
- [Background] Kendall PC, Flannery-Schroeder E, Panichelli-Mindel SM, Southam-Gerow M, Henin A, Warman M. Therapy for youths with anxiety disorders: a second randomized clinical trial. J Consult Clin Psychol. 1997 Jun;65(3):366-80. doi: 10.1037//0022-006x.65.3.366. PMID 9170760
- [Background] Kendall, P. C., & Hedtke, K. A. (2006). Cognitive-behavioral therapy for anxious children: Therapist manual (3rd ed.). Ardmore, PA: Workbook Publishing.
- [Background] Kendall PC, Hudson JL, Gosch E, Flannery-Schroeder E, Suveg C. Cognitive-behavioral therapy for anxiety disordered youth: a randomized clinical trial evaluating child and family modalities. J Consult Clin Psychol. 2008 Apr;76(2):282-97. doi: 10.1037/0022-006X.76.2.282. PMID 18377124
- [Background] Kolko DJ, Brent DA, Baugher M, Bridge J, Birmaher B. Cognitive and family therapies for adolescent depression: treatment specificity, mediation, and moderation. J Consult Clin Psychol. 2000 Aug;68(4):603-14. PMID 10965636
- [Background] Lejuez, C. W., Daughters, S. B., Danielson, C. W., & Ruggiero, K. (2006). The Behavioral Indicator of Resiliency to Distress (BIRD). Unpublished manual.
- [Background] Lewinsohn, P. M., Clarke,G.N., Hops, H., & Andrews, J. (1990). Cognitive-behavioral treatment for depressed adolescents. Behavior Therapy, 21, 385-401.
- [Background] Lewinsohn PM, Hops H, Roberts RE, Seeley JR, Andrews JA. Adolescent psychopathology: I. Prevalence and incidence of depression and other DSM-III-R disorders in high school students. J Abnorm Psychol. 1993 Feb;102(1):133-44. doi: 10.1037//0021-843x.102.1.133. PMID 8436689
- [Background] March, J. S. (1997). Multidimensional anxiety scale for children: Technical manual. North Tonawanda, NY: Multi-Health Systems, Inc.
- [Background] Moras K, Telfer LA, Barlow DH. Efficacy and specific effects data on new treatments: a case study strategy with mixed anxiety-depression. J Consult Clin Psychol. 1993 Jun;61(3):412-20. doi: 10.1037//0022-006x.61.3.412. PMID 8326041
- [Background] Muris, P. (2001) A brief questionnaire for measuring self-efficacy in youths. Journal of Psychopathology and Behavioral Assessment, 23(3), 145-149.
- [Background] Posner, K., Brent, D., Lucas, C., Gould, M., Stanley, B., Brown, G., ... & Mann, J. (2010). Columbia-Suicide Severity Rating Scale (C-SSRS): Pediatric/Cognitively Impaired - Lifetime Recent - Clinical. New York, NY: Research Foundation for Mental Hygiene, Inc.
- [Background] Poznanski, E. O., & Mokros, H.B. (1996). Manual for the Children's Depression Rating Scale-Revised. Los Angeles, CA: Western Psychological Services.
- [Background] Quinn, E. P., Brandon, T. H., & Copeland, A. L. (1996). Is task persistence related to smoking and substance abuse? The application of learned industriousness theory to addictive behaviors. Experimental and Clinical Psychopharmacology, 4(2), 186-190.
- [Background] Radloff, L.S. (1977). The CES-D Scale: a self-report depression scale for research in the general population. Applied Psychological Measures, 1, 385-401.
- [Background] Richards A, Richards LC, McGeeney A. Anxiety-related Stroop interference in adolescents. J Gen Psychol. 2000 Jul;127(3):327-33. doi: 10.1080/00221300009598587. PMID 10975428
- [Background] Ronan, K., Kendall, P. C., & Rowe, M. (1994). Negative affectivity in children: Development and validation of a questionnaire. Cognitive Therapy and Research, 18, 509-528.
- [Background] Rothbaum, F., Weisz, J. R., & Snyder, S. (1982). Changing the world and changing the self: A two-process model of perceived control. Journal of Personality and Social Psychology, 42, 5-37.
- [Background] Schniering CA, Rapee RM. Development and validation of a measure of children's automatic thoughts: the children's automatic thoughts scale. Behav Res Ther. 2002 Sep;40(9):1091-109. doi: 10.1016/s0005-7967(02)00022-0. PMID 12296494
- [Background] Shirk SR, Karver M. Prediction of treatment outcome from relationship variables in child and adolescent therapy: a meta-analytic review. J Consult Clin Psychol. 2003 Jun;71(3):452-64. doi: 10.1037/0022-006x.71.3.452. PMID 12795570
- [Background] Shirk, S., & Saiz, C. (1992). Clinical, empirical, and developmental perspectives on the therapeutic relationship in child psychotherapy. Development and Psychopathology, 4, 713-728.
- [Background] Silverman WK, Nelles WB. The Anxiety Disorders Interview Schedule for Children. J Am Acad Child Adolesc Psychiatry. 1988 Nov;27(6):772-8. doi: 10.1097/00004583-198811000-00019. No abstract available. PMID 3198566
- [Background] Silverman WK, Eisen AR. Age differences in the reliability of parent and child reports of child anxious symptomatology using a structured interview. J Am Acad Child Adolesc Psychiatry. 1992 Jan;31(1):117-24. doi: 10.1097/00004583-199201000-00018. PMID 1537762
- [Background] Silverman, W. K., & Albano, A. A. (1996). Anxiety Disorders Interview Schedule (ADIS-IV) Child and Parent Interview Schedules. US: Graywind Publications.
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. Motivation and Emotion, 29(2), 83-102.
- [Background] Solberg, M. E., & Olweus, D. (2003). Prevalence estimation of school bullying with the Olweus Bully/Victim Questionnaire. Aggressive Behavior, 29(3), 239-268.
- [Background] Spielberger, C. (1973). State-Trait Anxiety Interview for Children: Professional manual. Redwood City, CA: Mind Garden, Inc.
- [Background] Stark KD, Reynolds WM, Kaslow NJ. A comparison of the relative efficacy of self-control therapy and a behavioral problem-solving therapy for depression in children. J Abnorm Child Psychol. 1987 Mar;15(1):91-113. doi: 10.1007/BF00916468. PMID 3571741
- [Background] Stiffman AR, Horwitz SM, Hoagwood K, Compton W 3rd, Cottler L, Bean DL, Narrow WE, Weisz JR. The Service Assessment for Children and Adolescents (SACA): adult and child reports. J Am Acad Child Adolesc Psychiatry. 2000 Aug;39(8):1032-9. doi: 10.1097/00004583-200008000-00019. PMID 10939232
- [Background] Strauss, C. (1987). Modification of trait portion of State-Trait Anxiety Inventory for Children-parent form. (Available from the author, Department of Psychology, University of Florida, Gainesville, FL 32606)
- [Background] Strong D.R., Lejuez, C.W., Daughters S., Marinello M., Kahler C.W., & Brown, R.A. (2003) Unpublished manual. The computerized mirror tracing task, version 1.
- [Background] Stroop, J. (1935). Studies of interference in serial verbal reactions. Journal of Experimental Psychology, 28, 643-662.
- [Background] Temkin, A., B., Yadegar, M., Laurine, C. J., & Chu, B. C. Transdiagnostic approaches for children and adolescents. (In press). In T.H. Ollendick, S.W. White, & B.A. White (Eds.), The Oxford handbook of clinical child and adolescent psychology. London, UK: Oxford University Press.
- [Background] The Columbia Lighthouse Project/Center for Suicide Risk Assessment (2017). The Columbia Suicide Severity Rating Scale (C-SSRS): Supporting Evidence. Downloaded on 9/10/17 at: http://cssrs.columbia.edu/the-columbia-scale-c-ssrs/about-the-scale/
- [Background] Tottenham N, Tanaka JW, Leon AC, McCarry T, Nurse M, Hare TA, Marcus DJ, Westerlund A, Casey BJ, Nelson C. The NimStim set of facial expressions: judgments from untrained research participants. Psychiatry Res. 2009 Aug 15;168(3):242-9. doi: 10.1016/j.psychres.2008.05.006. Epub 2009 Jun 28. PMID 19564050
- [Background] Treadwell KR, Kendall PC. Self-talk in youth with anxiety disorders: states of mind, content specificity, and treatment outcome. J Consult Clin Psychol. 1996 Oct;64(5):941-50. doi: 10.1037//0022-006x.64.5.941. PMID 8916623
- [Background] Walkup JT, Albano AM, Piacentini J, Birmaher B, Compton SN, Sherrill JT, Ginsburg GS, Rynn MA, McCracken J, Waslick B, Iyengar S, March JS, Kendall PC. Cognitive behavioral therapy, sertraline, or a combination in childhood anxiety. N Engl J Med. 2008 Dec 25;359(26):2753-66. doi: 10.1056/NEJMoa0804633. Epub 2008 Oct 30. PMID 18974308
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Weersing VR, Weisz JR. Mechanisms of action in youth psychotherapy. J Child Psychol Psychiatry. 2002 Jan;43(1):3-29. doi: 10.1111/1469-7610.00002. PMID 11848335
- [Background] Weisz, J.R., Southam-Gerow, M.A., Gordis, E.B., & Connor-Smith, J. (2003). In A.E. Kazdin & J.R. Weisz (Eds.), Evidence-based Psychotherapies for Children and Adolescents (pp. 165-186). New York, NY: Guilford.
- [Background] Weisz JR, Thurber CA, Sweeney L, Proffitt VD, LeGagnoux GL. Brief treatment of mild-to-moderate child depression using primary and secondary control enhancement training. J Consult Clin Psychol. 1997 Aug;65(4):703-7. doi: 10.1037//0022-006x.65.4.703. PMID 9256573
- [Background] Weisz, J. R., Rothbaum, F. M., & Blackburn, T. F. (1984a). Standing out and standing in: The psychology of control in America and Japan. American Psychologist, 39, 955-969.
- [Background] Weisz, J. R., Rothbaum, F. M., & Blackburn, T. F. (1984b). Swapping recipes for control. American Psychologist, 39, 974-975.
- [Background] Weisz, J. R., Southam-Gerow, M. A., Gordis, E. B., & Connor-Smith, J. (2003). Primary and secondary control enhancement training for youth depression: Applying the deployment-focused model of treatment development and testing. In A. E. Kazdin & J. R. Weisz (Eds.), Evidence-based psychotherapies for children and adolescents (pp. 165-182). New York: Guilford Press.
- [Background] Weisz JR, Southam-Gerow MA, Gordis EB, Connor-Smith JK, Chu BC, Langer DA, McLeod BD, Jensen-Doss A, Updegraff A, Weiss B. Cognitive-behavioral therapy versus usual clinical care for youth depression: an initial test of transportability to community clinics and clinicians. J Consult Clin Psychol. 2009 Jun;77(3):383-96. doi: 10.1037/a0013877. PMID 19485581
- [Background] Weisz JR, Weiss B, Han SS, Granger DA, Morton T. Effects of psychotherapy with children and adolescents revisited: a meta-analysis of treatment outcome studies. Psychol Bull. 1995 May;117(3):450-68. doi: 10.1037/0033-2909.117.3.450. PMID 7777649
- [Background] Wood, J. J., Kiff, C. & Piacentini, J. C. (2005). Linkages among parental intrusiveness, dependency on caregivers at school, and separation anxiety in middle childhood. Manuscript in submission.
- [Background] Wechsler, D. (2003). Wechsler Intelligence Scale for Children-4th Edition. New York: Psychological Corporation.